CLINICAL TRIAL: NCT01414361
Title: Comparison of Fractional Flow Reserve (FFR) and Minimal Luminal Area (MLA) by Intravascular Ultrasound (IVUS) in Evaluating Intermediate Coronary Artery Stenosis: International Multi-center Study
Brief Title: Fractional Flow Reserve and Intravascular Ultrasound in Evaluating Intermediate Coronary Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Inje University (Other); Keimyung University (Other); Asan Medical Center (Other); Medstar Health Research Institute (Other); University of Florida (Other); National University of Singapore (Other)
Responsible Party: Division of cardiology / Cardiovascular center, Seoul National University Hospital
Other Study IDs: H-1106-077-366
Record Dates: First submitted 2011-08-09; First posted 2011-08-11 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Coronary Artery Stenosis
Keywords: Coronary artery stenosis; Fractional flow reserve; Intravascular ultrasonography
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intermediate lesion: intermediate lesions evaluated by both IVUS and FFR

SUMMARY:
Recent studies have shown that optimal IVUS criteria defining the functional significance (FFR < 0.8) of intermediate coronary stenoses is different according to their locations of the coronary tree. Herein, the investigators performed this study to validate these results and to generalize the IVUS criteria defining functional significance of intermediate coronary stenosis in a different location of coronary tree in a larger sample size.

DETAILED DESCRIPTION:
Both physiologic information from fractional flow reserve (FFR) and anatomical information from intravascular ultrasound (IVUS) in assessing intermediate coronary stenotic lesions are useful. Functional significance of a coronary stenosis is determined by both the severity of a stenosis and the amount of myocardium supplied. Therefore, when the functional significance of a lesion is assessed by lumen area measured by IVUS, different criteria should be applied according to lesion location and anatomical variations of the coronary artery. However, previous studies included only patients with proximal lesions or small vessel disease, and the sample sizes were too small to assess these differences. In a recent study, the investigators have shown that optimal IVUS criteria defining the functional significance (FFR < 0.8) of intermediate coronary stenoses is different according to their locations of the coronary tree. Herein, the investigators performed this study to validate the our results and to generalize the IVUS criteria defining functional significance of intermediate coronary stenosis in a different location of coronary tree in a larger sample size.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate coronary stenosis by visual estimation

Exclusion Criteria:

* history of coronary artery bypass graft surgery
* previously revascularized lesion
* creatinine > 1.6 mg/dL or eGFR < 30 ml/min/1.73m2 pre-procedure per institutional standards
* known pregnancy
* contrast agent allergy that cannot be adequately premedicated
* severe PVD precluding cardiac catheterization
* patient not a candidate for IVUS and FFR
* inability or unwillingness to provide informed consent
* inability or unwillingness to perform required follow up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate coronary stenosis who underwent both FFR and IVUS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
lumen area | day 1
  lumen area cut-off that can predict functional significance of a lesion

SECONDARY OUTCOMES:
angiographic stenosis, % plaque area | day 1
  angiographic and intravascular ultrasound parameters that can best predict the functional significance of lesions

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University
Locations (1):
- Seoul National University Hospital, Seoul, South Korea